CLINICAL TRIAL: NCT01221935
Title: A Retrospective Study To Evaluate The Current Utilization Of Desvenlafaxine Among Psychiatrists And Primary Care Physicians In The Treatment Of Patients With Major Depressive Disorder
Brief Title: Retrospective Study Evaluating The Current Utilization Of Desvenlafaxine Succinate Sustained-Release (Pristiq) Among Psychiatrists And Primary Care Physicians In The Treatment Of Patients With Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: 3151A1-4431; B2061039
Record Dates: First submitted 2010-10-13; First posted 2010-10-18 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Major Depressive Disorder
Keywords: retrospective chart review study; desvenlafaxine utilization; psychiatrists and primary care physicians; treatment of major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Serotonin and Noradrenaline Reuptake Inhibitors

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients initiated on Pristiq as a first line treatment
  Interventions: Other: Pristiq first-line treatment charts
- Patients initiated on Pristiq as a 2nd-line treatment
  Interventions: Other: Pristiq second-line treatment charts
- Patients initiated on a SNRI or SSRI as a first-line treatment
  Interventions: Other: SNRI or SSRI first-line treatment charts
- Patients initiated on a SNRI or SSRI as a 2nd-line treatment
  Interventions: Other: SNRI or SSRI second-line treatment charts

INTERVENTIONS:
Other: Pristiq first-line treatment charts — 300 charts including patients initiated on Pristiq within the past 6 months as a first-line treatment
  Groups: Patients initiated on Pristiq as a first line treatment
Other: Pristiq second-line treatment charts — 800 charts including patients initiated on Pristiq within the past 6 months as a second-line treatment (following first-line treatment with a Serotonin Norepinephrine Reuptake Inhibitor (SNRI) or Selective Serotonin Reuptake Inhibitors (SSRIs)).
  Groups: Patients initiated on Pristiq as a 2nd-line treatment
Other: SNRI or SSRI first-line treatment charts — 800 charts including patients initiated on a Serotonin Norepinephrine Reuptake Inhibitor (SNRI) or Selective Serotonin Reuptake Inhibitors (SSRIs) (excluding Pristiq) within the past 6 months as a first-line treatment.
  Groups: Patients initiated on a SNRI or SSRI as a first-line treatment
Other: SNRI or SSRI second-line treatment charts — 800 charts including patients initiated on a Serotonin Norepinephrine Reuptake Inhibitor (SNRI) or Selective Serotonin Reuptake Inhibitors (SSRIs)(excluding Pristiq) within the past 6 months as a second-line treatment (following the first-line treatment with a SNRI or SSRI).
  Groups: Patients initiated on a SNRI or SSRI as a 2nd-line treatment

SUMMARY:
The goal of this observational study is to learn about how Pristiq is currently being used in general practice and how psychiatrists and primary care physicians currently perceive Pristiq in terms of efficacy, tolerability, and adherence compared to other treatments for major depressive disorder (MDD).

DETAILED DESCRIPTION:
It is retrospective patient chart study among psychiatrists and primary care physicians (PCPs) treating patients suffering from major depressive disorder (MDD). Physicians will be asked general medical questions in order to quantify their prescribing behavior and their perception of treatment performance. A retrospective patient chart review will then be performed and patient data will be collected to document patient characteristics and actual treatment outcomes. Upon qualification, specific instructions for chart review will be provided. Once the identified charts are pulled, the physicians are instructed to continue with the on-line survey. In total, there will be approximately 450 psychiatrists and 450 primary care physicians participating in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be adult, diagnosed with major depressive disorder and treated with pharmacotherapy.
* Physicians must be either a psychiatrist or a primary care physician, a prescriber of Pristiq, have at least 3 charts representing the 4 identified patient types, have been in clinical practice between 4 and 35 years, primarily office based (50%+), not participated in a research study relating to antidepressants or antidepressant therapy within the past month, not a consultant or have a professional relationship with a pharmaceutical company other than for clinical trials or speaking engagements, and not be employed by of affiliated with an advertising agency, market research company, or pharmaceutical company.

Exclusion Criteria:

* Patients who have not been treated for depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient charts from psychiatrists and primary care physicians (PCPs) treating patients suffering from major depressive disorder (MDD).
Sampling Method: Non-Probability Sample
Enrollment: 2701 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
300 charts including patients initiated on Pristiq within the past 6 months as a first-line treatment. | 6 months
800 charts including patients initiated on Pristiq within the past 6 months as a second-line treatment (following first-line treatment with a SNRI or SSRI). | 6 months
800 charts including patients initiated on a SNRI or SSRI (excluding Pristiq) within the past 6 months as a first-line treatment. | 6 months
800 charts including patients initiated on a SNRI or SSRI (excluding Pristiq) within the past 6 months as a second-line treatment (following the first-line treatment with a SNRI or SSRI). | 6 months

SECONDARY OUTCOMES:
Incidence of adverse events and Incidence of discontinuation due to adverse events | 6 months
Percent of patients experiencing relapse | 6 months
Length of time to relapse | 6 months
Percent of discontinuation / medication switches due to lack of efficacy | 6 months
Subjective physician assessment of symptom control | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-4431&StudyName=Retrospective%20Study%20Evaluating%20The%20Current%20Utilization%20Of%20Desvenlafaxine%20Succinate%20Sustained-Release%20%28Pristiq%29%20Among%20Pychiatrists%20And%20Prima